CLINICAL TRIAL: NCT00140192
Title: Creatine as a New Treatment for Schizophrenia:A Double-Blind Trial
Brief Title: Creatine Treatment in Psychiatric Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BMHC-3835
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2005-10

CONDITIONS: Schizophrenia
Keywords: creatine metabolism; schizophrenia; energy metabolism
MeSH Terms: conditions — Schizophrenia | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: creatine

SUMMARY:
Creatine plays a pivotal role in brain energy homeostasis. Creatine supplementation is widely used in enhancing sports performance, and has been tried in the treatment of neurological, neuromuscular and atherosclerotic disease with a paucity of side effects.

Dechent et al (1999) studied the effect of oral creatine supplementation for 4 wk demonstrating a statistically significant increase of mean concentration of total creatine across brain regions. These findings suggest the possibility of using oral creatine supplementation to modify brain high-energy phosphate metabolism in subjects with various brain disorders, including schizophrenia and major depression. Recently, Rae et al (2003) reported that creatine supplementation for 6 weeks had a significant positive effect on both working memory and Raven matrices. Several independent lines of evidence suggest the possible involvement of altered cerebral energy metabolism in schizophrenia.

We are performing a double blind cross-over study of creatine in schizophrenia.

Forty patients will be treated with creatine for 3 months in a double-blind crossover design. Rating scales will include scales for assessing negative and positive symptoms of schizophrenia, clinical global impressions scale, scales for side-effects and a cognitive battery

Creatine effects on brain energy metabolism and its possible cognitive enhancing properties raise the possibility of developing a new therapeutic strategy in schizophrenia focusing on treating metabolic hypoactive brain areas including frontal regions.

DETAILED DESCRIPTION:
Creatine plays a pivotal role in brain energy homeostasis, being a temporal and spatial buffer for cytosolic and mitochondrial pools of the cellular energy currency adenosine triphosphate (Wyss & Kaddurah-Daouk, 2000). Recent studies have suggested increased brain utilization of oxygen following oral creatine supplementation (Persky & Brazeua, 2001). Creatine supplementation is widely used in enhancing sports performance, and has been tried in the treatment of neurological, neuromuscular and atherosclerotic disease with a paucity of side effects (Persky & Brazeua, 2001).

Creatine enters the brain via a specialized sodium dependent transporter. Dechent et al (1999) studied the effect of oral creatine supplementation of 20g/day for 4 wk demonstrating a significant increase of mean concentration of total creatine across brain regions (8.7% corresponding to 0.6mM, P < 0.001). Lyoo et al (2003) studied magnetic resonance spectroscopy of high-energy phosphate metabolites in human brain following oral supplementation of creatine reporting that creatine (0.3 g/kg/day for the first 7 days and 0.03 g/kg/day for the next 7 days) significantly increased brain creatine levels. These findings suggest the possibility of using oral creatine supplementation to modify brain high-energy phosphate metabolism in subjects with various brain disorders, including schizophrenia and major depression, where alterations in brain high-energy phosphate metabolism have been reported.

Kieburtz et al (see: http://www.huntington-study-group.org/Creatine%20abstract.htm) are conducting a double blind clinical trial of creatine in 50 ambulatory Huntington disease subjects randomized to creatine or placebo. Those randomized to creatine receive 3g for 2 months and then 5g for an additional 2 months. There have been no significant adverse events associated with creatine or significant changes in laboratory tests or vital signs. In the creatine treated group creatine plasma levels approximately doubled (210 ± 335 µM vs. 500 ± 125 µM). Kieburtz et al are currently also conducting a multi-center, double-blind study of creatine in patients with Parkinson's disease, funded by the National Institute of Neurological Disorders and Stroke (NINDS). Recently, Rae et al (2003) reported that creatine supplementation (5 grams per day for 6 weeks) had a significant positive effect (p < 0.0001) on both working memory (backward digit span) and Raven's Advanced Progressive Matrices. These findings suggest a role of brain energy capacity in influencing brain cognitive performance and that creatine via its effects on brain energy metabolism may exert beneficial effects on cognition.

Several independent lines of evidence suggest the possible involvement of altered cerebral energy metabolism in the pathophysiology of schizophrenia. Imaging studies have used positron emission tomography (PET) with flurodeoxyglucose (FDG), or functional magnetic resonance imaging (fMRI), 15O magnetic resonance spectroscopy with 31P (31P-MRS) and single photon emission tomography (SPECT), to investigate cerebral metabolic rates in schizophrenia. Most but not all studies reveal decreased metabolism in the frontal cortex in schizophrenia, which was termed hypofrontality. Several studies also observed alterations in brain metabolic rates in other brain regions including the temporal lobes, the thalamus and the basal ganglia, leading to the suggestion of an impairment in the fronto-striatal-thalamic circuitry in schizophrenia rather than in a specific brain region (Andreasen et al. 1997). A direct link to phosphocreatine and ATP energy systems came from studies using 31P-MRS with or without chemical shift imaging, which enabled the measurement of ATP, phosphocreatine and inorganic phosphate. These studies showed reduced ATP in the frontal lobe and in left temporal lobe of schizophrenic patients as compared to controls (Volz et al. 2000). Altered brain energy metabolism could be due to impairment of mitochondria and a variety of studies reviewed recently by Ben Shachar (2002) suggest impaired mitochondrial energy metabolism in schizophrenia.

Interestingly, creatine besides its energy sparing properties was also shown to have neuroprotective properties in a variety of animal models for brain diseases including Huntington and Parkinson diseases, as well as exerting protective effects in animal models for cerebral hypoxia (Persky & Brazeua, 2001).

We are performing a double blind cross-over study of creatine in schizophrenia.

Forty consenting schizophrenic patients, 18-60 years old, physically healthy, with more than 2 years of illness in a stable condition (no gross changes in clinical presentation in the last 6 months as judged by the patient's psychiatrist) and presenting negative and cognitive symptoms (as judged by the patient's psychiatrist along with score in at least 3 items of the PANSS negative subscale =4 points, while items of the PANSS positive subscale scored = 3 points). These patients will be recruited into the study over two years.

Excluded will be patients with alcohol or drug abuse in the 6 months prior to entry into the study or any clinically significant medical condition or laboratory abnormality.

Twenty patients will be treated with creatine for 3 months (3 g daily in the first month and then 5 g daily for another 2 months) and then for 3 months with placebo. The other twenty patients will be administered placebo for 3 months and then creatine for 3 months in the same dosages and procedure. Patients' neuroleptic treatment will not be affected by study participation. Mood stabilizers, benzodiazepines and anticholinergic medications are allowed but doses will be documented throughout the study. Routine blood tests including kidney function, liver function as well as plasma creatine and creatinine will be monitored at baseline and monthly throughout the study.

Positive and Negative Syndrome Scale (PANSS), Clinical Global Impressions (CGI), and Adverse effect/side effects assessment will be administered at baseline and then monthly. A Cognitive Battery will be administered at baseline, three months, and six months consisting of the California Verbal Learning Test; Trail making A&B; Purdue Pegboard; Digit Symbol Coding; Continuous performance test ; Reaction Time performance Test and Wisconsin Card Sort Test.

Power Analysis: We have demonstrated significant effects as add-on in schizophrenia in this design with folate treatment as a homocysteine lowering strategy in schizophrenia. A sample of 36 subjects recruited over 24 months showed a statistically significant, clinically relevant difference between the active treatment and placebo in a similar design to that proposed here.

Creatine administration is safe with a paucity of side effects. Creatine effects on brain energy metabolism and its possible cognitive enhancing properties raise the possibility of developing a new therapeutic strategy in schizophrenia focusing on treating metabolic and energetic hypoactive brain areas including frontal regions. My personal research experience and position at the Beersheva Mental Health Centre make such a trial eminently feasible.

REFERENCES

Andreasen NC, O'Leary DS, Flaum M, Nopoulos P, Watkins GL, Boles Ponto LL, et al. Hypofrontality in schizophrenia: distributed dysfunctional circuits in neuroleptic-naive patients. Lancet 1997; 349: 1730-4.

Ben-Shachar D. Mitochondrial dysfunction in schizophrenia: a possible linkage to dopamine. J Neurochem 2002; 83: 1241-51.

Dechent P, Pouwels PJ, Wilken B, Hanefeld F, Frahm J. Increase of total creatine in human brain after oral supplementation of creatine-monohydrate. Am J Physiol 1999; 277: R698-704.

Lyoo IK, Kong SW, Sung SM, Hirashima F, Parow A, Hennen J, et al. Multinuclear magnetic resonance spectroscopy of high-energy phosphate metabolites in human brain following oral supplementation of creatine-monohydrate. Psychiatry Res 2003; 123: 87-100.

Persky AM, Brazeau GA. Clinical pharmacology of the dietary supplement creatine monohydrate. Pharmacol Rev 2001; 53: 161-76.

Rae C, Digney AL, McEwan SR, Bates TC. Oral creatine monohydrate supplementation improves brain performance: a double-blind, placebo-controlled, cross-over trial. Proc R Soc Lond B Biol Sci 2003; 270: 2147-50.

Volz H, Gaser C, Sauer H. Supporting evidence for the model of cognitive dysmetria in schizophrenia--a structural magnetic resonance imaging study using deformation-based morphometry. Schizophr Res 2000; 46: 45-56.

Wyss M, Kaddurah-Daouk R. Creatine and creatinine metabolism. Physiol Rev 2000; 80: 1107-213.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60
* physically healthy
* at least 2 years of illness in a stable condition
* presenting negative and cognitive symptoms

Exclusion Criteria:

* drug or alcohol abuse
* clinically significant medical condition
* laboratory abnormality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2004-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale
Clincal Global Impression

CONTACTS AND LOCATIONS:
Overall Officials: RH Belmaker, MD, Study Director — Ben Gurion University of the Negev + Beersheva Mental Health Center
Locations (1):
- Beersheva Mental Health Center, Beersheva, Israel

REFERENCES:
- [Derived] Kaptsan A, Odessky A, Osher Y, Levine J. Lack of efficacy of 5 grams daily of creatine in schizophrenia: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2007 Jun;68(6):881-4. doi: 10.4088/jcp.v68n0609. PMID 17592912